CLINICAL TRIAL: NCT05509153
Title: A Randomised Controlled Trial, Of N-Acetyl Cysteine (NAC), for Premanifest Huntingtin Gene Expansion Carriers
Acronym: NAC-preHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Collaborators: Deakin University (Other); Monash University (Other); Royal Perth Hospital (Other); The University of Queensland (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Clement Loy, Director and Neurologist, Huntington Disease Service, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/ETH12013
Record Dates: First submitted 2022-08-08; First posted 2022-08-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Huntington Disease
Keywords: N-Acetylcysteine
MeSH Terms: conditions — Huntington Disease | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either the NAC arm or the placebo arm using Block Randomisation, stratified by site, through a centralised process, with allocation concealment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC (Experimental): 1g N-Acetylcysteine capsules, taken orally twice a day.
  Interventions: Drug: NAC
- Placebo (Placebo Comparator): Coated Placebo capsules, taken orally twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAC — 1g of clinical grade N-Acetylcysteine capsules, taken orally twice a day
  Other Names: N-Acetylcysteine
  Arms: NAC
Drug: Placebo — Coated Placebo capsules, manufactured to match appearance and taste, taken orally twice a day
  Arms: Placebo

SUMMARY:
NAC-preHD is a phase II randomized placebo controlled study of oral NAC among premanifest HD gene expansion carriers, with clinical and radiological outcome at three years.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Huntingtin gene expansion carrier with >= 39 CAG repeats
* Absence of unequivocal motor signs of HD - that is, UHDRS
* Diagnostic Confidence Level needs to be <4 upon enrolment
* Expected to develop clinical HD within 10 years of trial enrolment using the Langbehn formula
* Availability of an informant for corroborative history
* Negative serum pregnancy test for women of childbearing potential
* If of childbearing potential, is able and agrees to remain abstinent or use adequate contraceptive methods
* Ability to tolerate MRI scans
* Ability to tolerate blood draws
* Able to comply with all study protocol requirements, according to the investigators judgement
* In the opinion of the investigator, medically, psychiatrically and neurologically stable at the time of enrolment

Exclusion Criteria:

* Diagnosis of clinical HD
* Known hypersensitivity to NAC
* Pregnancy, breastfeeding or intention to do so prior to the end of the study
* Exposure to any investigational drugs within 30 days of Baseline Visit
* Use of supplemental NAC
* Abnormalities in laboratory measurements, ECG or vital signs at screening, which precludes safe participation in the study
* Current or history of substance abuse within one year of Baseline visit
* Unstable psychiatric or acute medical illness including cancer, as determined by investigator
* Current use of antipsychotic medications or Tetrabenazine
* History of gene therapy, cell transplantation, or any experimental brain surgery
* History of attempted suicide or suicidal ideation within 12 months prior to screening
* Pre-existing structural brain lesion as assessed by a centrally read MRI scan during the screening period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Caudate Atrophy Rate on volumetric MRI | Baseline through end of study (up to 3 years)
  Blinded assessment
Rate of motor phenoconversion | Baseline through end of study (up to 3 years)
  Defined by conversion to Diagnostic Confidence Level 4, upon blinded assessment using the UHDRS motor subscale

SECONDARY OUTCOMES:
UHDRS motor subscale (total score) | Baseline through end of study (up to 3 years)
  Measuring changes in motor function
Stroop Word | Baseline through end of study (up to 3 years)
  Change in cognition as measured by Stroop Word
Trail Making Test | Baseline through end study (up to 3 years)
  Change in cognition as measured by Trail Making Test
Montreal Cognitive Assessment | Baseline through end of study (up to 3 years)
  Change in cognition as measured by Montreal Cognitive Assessment
Symbol Digit Modality Test | Baseline through end of study (up to 3 years)
  Change in cognition as measured by Symbol Digit Modality Test
Changes in Mood and Behavioural symptoms | Baseline through end of study (up to 3 years)
  Evaluated using the PBA-s, a semi-structured interview behavioural scale
Changes in Daily Function | Baseline through end of study (up to 3 years)
  Measured using the Total Functional Capacity and Independent Scale from the broader UHDRS and the Functional Rating Scale for HD
Change to Quality of Life | Baseline through end of study (up to 3 years)
  As measured by the standardised questionnaires, HDQoL and EQ-5D
Study completion (Safety and Tolerability) | Baseline through end of study (up to 3 years)
  Measured by the proportion of participants completing NAC arm of study
Incidence of abnormal laboratory values and/or 12-lead ECG changes (Safety and Tolerability) | Baseline through end of study (up to 3 years)
  Measured by the Number of participants with abnormal laboratory values and/or 12-lead ECG changes compared to baseline
Incidence of adverse and/or serious adverse events (Safety and Tolerability) | Baseline through end of study (up to 3 years)
  Measured by the number of adverse and/or serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clement Loy, Principal Investigator — University of Sydney; Yenni Lie, Principal Investigator — Calvary Health Care Bethlehem; Dennis Velakoulis, Principal Investigator — Melbourne Health; Carolyn Orr, Principal Investigator — Perron Institute; John O'Sullivan, Principal Investigator — The University of Queensland; Rob Adam, Principal Investigator — The University of Queensland
Locations (5):
- Australia (5):
  - Westmead Hospital, Westmead, New South Wales
  - The University of Queensland, Herston, Queensland
  - Calvary Health Care Bethlehem, Parkdale, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Perron Institute, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided
Currently not included in ethics approval but to be investigated.